CLINICAL TRIAL: NCT05916768
Title: Management of Acute Bronchitis in Switzerland With Pelargonium Sidoides Extract EPs®7630 Versus Usual Care - a Pragmatic, Open-label, Randomised Controlled Trial
Brief Title: Management of Acute Bronchitis With Pelargonium Sidoides Extract
Acronym: Phytobronch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Fribourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00125
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Bronchitis
Keywords: pelargonium sidoides
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The solution of Pelargonium sidoides extract EPs® 7630:
  3x30 drops/day for 7 days and will be advised to pursue the treatment until the end of symptoms if bothered by the cough up to a maximum of 21 days.
  Interventions: Other: Pelargonium sidoides extract EPs® 7630
- Control group (Active Comparator): Usual care. Reference therapies, which are classified as symptomatic treatments, are chosen freely by the PCP except for phytotherapy
  Interventions: Other: usual care

INTERVENTIONS:
Other: Pelargonium sidoides extract EPs® 7630 — Kaloba® solution, a standardized alcoholic extract obtained from the roots of Pelargonium sidoides (EPs® 7630).
  Arms: Intervention group
Other: usual care — symptomatic treatments
  Arms: Control group

SUMMARY:
The aim of our study is to conduct a pragmatic RCT meeting all required standards to evaluate the effectiveness of Pelargonium sidoides extract, EPs® 7630, in the management of acute bronchitis with or without COVID-19 in PCP practices and walk-in clinics in French-speaking Switzerland. The RCT will be preceded by a pilot phase to ensure its feasibility.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effectiveness of Pelargonium sidoides extract EPs® 7630, also known under the brand name Kaloba®, in the management of acute bronchitis.

The main questions it aims to answer are:

* Is Pelargonium sidoides extract EPs® 7630 effective to reduce the severity and the duration of symptoms related to acute bronchitis ?
* Does Pelargonium sidoides extract EPs® 7630 allow to reduce the prescription of antibiotics?

Participants will be randomize 1:1 either in the control group (usual care) or in the intervention group (Pelargonium sidoides extract EPs® 7630).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 and over) consulting for the first time, for the same episode, either for an acute cough (≤8 days) as the main symptom, suggestive of acute bronchitis, or for an illness (≤8 days) in which cough is not the main symptom but PCP believes that acute bronchitis is the most likely diagnosis.
* Patients tested positive to COVID-19 who meet the above-mentioned criteria will be included too.

Exclusion Criteria:

* Infection requiring antibiotic treatment (ex. cystic fibrosis)
* Pneumonia
* Known hypersensitivity to Pelargonium sidoides extract or excipients of the trial medication
* Non-infectious causes (COPD, asthma, pulmonary embolism, heart failure, gastroesophageal reflux, allergy)
* Lacking the faculty of discernment (for example: dementia, decompensated psychosis or severe depression)
* Inability to fill out the diary (no ability to read and understand French)
* Pregnancy or breastfeeding
* Immunological deficiencies
* Hospitalization
* Severe hepatic disease
* Patients who have already started a treatment with Pelargonium sidoides EPs® 7630 for this current episode (Kaloba®, Umckaloabo®)
* Important risk of bleeding (severe thrombocytopenia and anticoagulant intake)
* If the patient is taking a drug among these classes of drugs:

anticoagulants, immunosuppressants, chemotherapy or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Pelargonium sidoides extract EPs® 7630 | 22 days
  Effectiveness will be determined by comparing the number of days needed to achieve a 50% reduction in the ABSS score after peak of symptoms in each group.
Proportion of patients taking antibiotics | 22 days
  The co-medication, including antibiotics, will be collected by the investigator at day 4, 8 and 22. The results will be compared between the two arms.

SECONDARY OUTCOMES:
Integration of a herbal medicinal product in conventional settings | 22 days
  Proportion of primary care physicians (PCPs) who agreed to participate in the study

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Rodondi, Prof., Principal Investigator — University of Fribourg
Locations (1):
- University of Fribourg, Fribourg, Canton of Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No
anonymised database, only for patients who signed the consent statement for the re-use of data in coded form.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT05916768/Prot_SAP_000.pdf